CLINICAL TRIAL: NCT04327232
Title: Mineralocorticoid Antagonism to Stop Progression of Atrial Fibrillation (MONITOR-AF) Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: University of Otago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Monitor-AF
Record Dates: First submitted 2019-06-12; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): For patients randomized to active experimental arm: Spironolactone
  Patient will receive study drug for 18 months. Study drug dosages are 1 tablet alternate day, 1 tablet per day, or 2 tablets per day, with 1 tablet being 25mg spironolactone. Study drugs are titrated every 3 months based on patients' potassium and eGFR blood tests results.
  Interventions: Drug: Spironolactone 25mg
- Control (Placebo Comparator): For patients randomized to control arm: Placebo
  Patient will receive placebo for 18 months. Placebo dosages are 1 tablet alternate day, 1 tablet per day, or 2 tablets per day. Placebo are titrated every 3 months based on patients' potassium and eGFR blood tests results.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Spironolactone 25mg — Mineralocorticoid Receptor Antagonists
  Arms: Active
Drug: Placebo oral tablet — Placebo
  Arms: Control

SUMMARY:
This proposal details the implementation of an international (Singapore and New Zealand) multi-centre study to test a novel therapeutic strategy aimed at reducing the burden of atrial fibrillation - an important medical condition with major healthcare implications. Unique aspects of this study include i) a non-arrhythmic treatment target (mineralocorticoid receptor antagonism) -targeting the arrhythmogenic substrate of AF before it becomes permanently established, ii) the use of pacemaker monitoring capability to accurately document AF burden, thus increasing the power of the study and iii) multi-national collaborative, double blind design.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years (without child-bearing potential for women);
* With a permanent pacemaker capable of AF monitoring;
* Device documented AF in the last 12 months; Defined as:

  i. atrial high rate events (AHRE) > 220 bpm for >1% of the time; or ii. > 6 mins on at least one occasion

Exclusion Criteria:

* Persistent (defined as sustained AF lasting continuously for 7 or more days)
* History of heart failure with indication for MRAs
* Any existing clinical indication for MRA or K+ sparing diuretic such as uncontrolled hypertension or oedema
* Contraindication to MRA
* Severe renal dysfunction (eGFR <30ml/min by CKD-Epi)
* Sustained hyperkalaemia (defined as K+ >5mmol/L in the absence of reversible cause)
* Receiving AF suppression pacing
* Women of child bearing potential
* Patients taking medications which may interact with the study drug or increase the level of potassium in the blood, include lithium, amiloride, cyclosporine, eplerenone, tacrolimus, and triamterene.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Development of persistent AF (defined as the first episode of sustained AF lasting for more than 7 days) | 18 months
  Development of persistent AF (defined as the first episode of sustained AF lasting for more than 7 days)

SECONDARY OUTCOMES:
Percentage of total time in AF. | 18 months
  Percentage of total time in AF.
Number of AF episodes | 18 months
  Number of AF episodes > 5 minutes duration recorded on pacemaker
Number of symptomatic AF episodes | 18 months
  Number of symptomatic AF episodes
Number of admissions for AF | 18 months
  Number of admissions for AF
Change in LA volumes in millimetre | 18 months
  Change in LA volumes in millimetre assessed by echo scan
Change in LV volumes in millimetre | 18 months
  Change in LV volumes in millimetre assessed by echo scan
Change in systolic and diastolic function | 18 months
  Change in systolic and diastolic function assessed by echo scan
Change in cardiac and systemic markers | 18 months
  Change in cardiac and systemic markers of stretch assessed by biomarkers blood tests - NT-proBNP
Change in cardiac and systemic markers of inflammation | 18 months
  Change in cardiac and systemic markers of inflammation assessed by biomarkers blood tests - hsCRP, myeloperoxidase, ST-2, GD-15, Galectin-3
Change in cardiac and systemic markers of fibrosis | 18 months
  Change in cardiac and systemic markers of fibrosis assessed by biomarkers blood tests - PIIP, type 1 and II procollagen

CONTACTS AND LOCATIONS:
Locations (4):
- Singapore (4):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore